CLINICAL TRIAL: NCT01313650
Title: A 24-Week, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GSK573719/GW642444 Inhalation Powder and the Individual Components Delivered Once-Daily Via a Novel Dry Powder Inhaler in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 24-week Evaluation of GSK573719/Vilanterol (62.5/25mcg) and Components in COPD
Acronym: DB2113373
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113373; 2010-023349-32 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: long-acting beta agonist; anticholinergic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK573719/GW642444 (Experimental): 62.5/25mcg
  Interventions: Drug: 62.5/25mcg
- GSK573719 (Experimental): 62.5mcg
  Interventions: Drug: 62.5mcg
- GW642444 (Experimental): 25mcg
  Interventions: Drug: 25mcg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 62.5/25mcg — GSK573719/GW64244
  Arms: GSK573719/GW642444
Drug: 62.5mcg — GSK573719
  Arms: GSK573719
Drug: 25mcg — GW642444
  Arms: GW642444
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase III multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of GSK573719/GW642444 Inhalation Powder, GSK573719 Inhalation Powder, GW642444 Inhalation Powder and Placebo when administered once-daily via a Novel Dry Powder Inhaler over a 24-week treatment period in subjects with COPD. Subjects who meet eligibility criteria at Screening (Visit 1) will complete a 7 to14 day run-in period followed by a randomization visit (Visit 2) then a 24-week treatment period. There will be a total of 9 clinic study visits. A follow-up phone contact for adverse event assessment will be conducted approximately one week after the last study visit (Visit 9 or Early Withdrawal). The total duration of subject participation in the study will be approximately 27 weeks. A subset of subjects at selected sites will also perform 24-hour serial spirometry and Holter monitoring during the study and provide serial blood samples for pharmacokinetic analysis. Sparse pharmacokinetic sampling for population pharmacokinetic analyses will be obtained from non-subset subjects. The primary measure of efficacy is clinic visit trough (pre-bronchodilator and pre-dose) FEV1 on Treatment Day 169. Safety will be assessed by adverse events, 12-lead ECGs, vital signs, clinical laboratory tests, and 24 hour Holter monitoring (subset only).

DETAILED DESCRIPTION:
This is a 24-week, phase III multicenter, randomized, double-blind, placebo-controlled, parallel-group study.

Eligible subjects will be randomized to GSK573719/GW642444 125/25mcg, GSK573719 125mcg, GW642444 25mcg, and placebo treatment groups in a 3:3:3:2 ratio such that of the planned 1463 total number of randomized subjects approximately 399 subjects will be randomized to each active treatment group and 266 subjects will be randomized to placebo. All treatments will be administered once-daily in the morning by inhalation using a Novel Dry Powder Inhaler (Novel DPI).

There will be a total of 9 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 7 to 14 day run-in period followed by a 24-week treatment period. Clinic visits will be at Screening, Randomization (Day 1), Day 2, after 4, 8, 12, 16, and 24-weeks of treatment, and 1 day after the Week 24 Visit (also referred as Treatment Day 169). A follow-up contact for adverse assessment will be conducted by telephone approximately 7 days after Visit 9 or the Early Withdrawal Visit. The total duration of subject participation, including follow-up will be approximately 27 weeks. All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the run-in and study treatment periods.

At screening, pre-bronchodilator spirometry testing will be followed by post-albuterol/salbutamol spirometry testing. Post-albuterol/salbutamol FEV1 and FEV1/FVC values will be used to determine subject eligibility. To further characterize bronchodilator responsiveness, post-ipratropium testing will be conducted following completion of post-albuterol/salbutamol spirometry.

Spirometry will be conducted at each post-randomization clinic visit. Six hour post-dose serial spirometry will be conducted at Visits 2, 4, 6, and 8. Trough spirometry will be obtained 23 and 24 hours after the previous day's dose of blinded study medication at Visits 3 to 9. All subjects will be provided with an electronic diary (eDiary) for completion daily in the evening throughout the run-in and treatment periods. Subjects will use the eDiary to record dyspnea scores using the Shortness of Breath with Daily Activities instrument (SOBDA), daily use of supplemental albuterol/salbutamol as either puffs/day from a metered-dose inhaler (MDI) and/or nebules used per day, and any healthcare contacts related to COPD.

Additional assessments of dyspnea will be obtained using the Baseline and Transition Dyspnea Index (BDI/TDI) which is an interviewer based instrument. At Visit 2, the severity of dyspnea at baseline will be assessed using the BDI. At subsequent visits (Visits 4, 6, and 8) change from baseline will be assessed using the TDI. Disease specific health status will be evaluated using the subject-completed St. George's Respiratory Questionnaire (SGRQ). The SGRQ will be completed at Visits 2, 4, 6, and 8. Administration of the SGRQ and BDI/TDI should be done prior to spirometry testing.

The occurrence of adverse events will be evaluated throughout the study beginning at Visit 2. SAEs will be collected over the same time period as for AEs. However, any SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded from the time a subject consents to participate in the study up to and including any follow up contact.

Additional safety assessments of vital signs (blood pressure and pulse rate), 12-lead ECGs and standard clinical laboratory tests (hematology and chemistry) will be obtained at selected clinic visits. Blood samples for population pharmacokinetic analyses will be obtained.

At selected study sites, a subset of approximately 198 subjects will perform 24-hour serial spirometry during the study for evaluation of lung function over the dosing period. In conjunction with the serial spirometry, this subset of subjects will also perform 24 hour Holter monitoring and provide blood samples for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* 10 pack-year or greater history of cigarette smoking
* Post-bronchodilator FEV1/FVC of <0.7
* Predicted FEV1 of 70% of normal or less
* Modified Medical Research Council (mMRC) dyspnea score of 2 or greater

Exclusion Criteria:

* Women who are pregnant, lactating, or planning to become pregnant
* Respiratory disorders other than COPD, including a current diagnosis of asthma
* Clinically significant non-respiratory diseases or abnormalities that are not adequate controlled
* Significant allergy or hypersensitivity to anticholinergics, beta-agonist, or the excipients of magnesium stereate or lactose used in the inhaler delivery device
* Hospitalization for COPD or pneumonia within 12 weeks prior to screening
* Lung volume reduction surgery within 12 weeks prior to screening
* Abnormal and clinically significant ECG findings at screening
* Clinically significant laboratory findings at screening
* Use of systemic corticosteroids, antibiotics for respiratory tract infections, strong cytochrome P450 3A4 inhibitors, high dose inhaled steroids (>1000mcg fluticasone propionate or equivalent), PDE4 inhibitors, tiotropium, oral beta2-agoinists, short- and long-acting inhaled beta2-agonists, ipratropium, inhaled sodium cromoglycate or nedocromil sodium, or investigational medicines for defined time periods prior to the screening visit
* Use of long-term oxygen therapy (12 hours or greater per day)
* Regular use of nebulized treatment with short-acting bronchodilators
* Participation in the acute phase of a pulmonary rehabilitation program
* A know or suspected history of alcohol or drug abuse
* Affiliation with the investigational site
* Previous use of GSK573719 or GW642444 alone or in combination, including the combination of fluticasone furoate and GW64244

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1538 (Actual)
Dates: Start 2011-03-01; Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (144):
- United States (36):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Olathe, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Larchmont, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Phoenixville, Pennsylvania
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Pelzer, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Bulgaria (7):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Troyan Municipality
  - GSK Investigational Site, Varna
- Canada (11):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (6):
  - GSK Investigational Site, Rancagua, Reg Del Libert Bern Ohiggins
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talcahuano
  - GSK Investigational Site, Viña del Mar
- Czechia (11):
  - GSK Investigational Site, Český Krumlov
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Kyjov
  - GSK Investigational Site, Lovosice
  - GSK Investigational Site, Nový Jičín
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Praha 5 - Radotin
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Teplice
- Greece (6):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari / Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Serres
  - GSK Investigational Site, Thessaloniki
- Japan (10):
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Puebla, Pue, Puebla
- Poland (10):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gidle
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Iława
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Łomża
- Russia (14):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl
- South Africa (9):
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Meyerspark, Gauteng
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Newtown
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Tygerberg
- Spain (15):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Badalona / Barcelona
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Salt (gerona)
  - GSK Investigational Site, Sant Boi de Llobregat - Barcelona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- Thailand (5):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Nonthaburi
  - GSK Investigational Site, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Donohue JF, Maleki-Yazdi MR, Kilbride S, Mehta R, Kalberg C, Church A. Efficacy and safety of once-daily umeclidinium/vilanterol 62.5/25 mcg in COPD. Respir Med. 2013 Oct;107(10):1538-46. doi: 10.1016/j.rmed.2013.06.001. Epub 2013 Jul 2. PMID 23830094
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113373 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria at Screening (Visit 1) completed a 7 to 10-day run-in period and were then randomized to a 24-week treatment (trt.) period. A total of 2210 participants were screened; 1536 participants were randomized and 1532 participants took at least one dose of randomized medication.
Groups:
- Placebo: Participants received matching placebo once daily (QD) via a dry powder inhaler (DPI) in the morning for 24 weeks.
- UMEC 62.5 µg QD: Participants received umeclidinium bromide (UMEC) 62.5 micrograms (µg) QD via a DPI in the morning for 24 weeks.
- VI 25 µg QD: Participants received vilanterol (VI) 25 µg QD via a DPI for 24 weeks.
- UMEC/VI 62.5/25 µg QD: Participants received UMEC/VI 62.5/25 µg QD via a DPI in the morning for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD
Started | 280 | 418 | 421 | 413
Completed | 204 | 324 | 318 | 332
Not Completed | 76 | 94 | 103 | 81
Not completed — Adverse Event | 9 | 34 | 24 | 23
Not completed — Lack of Efficacy | 37 | 20 | 32 | 20
Not completed — Lost to Follow-up | 1 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 16 | 20 | 15 | 15
Not completed — Protocol Violation | 4 | 7 | 5 | 6
Not completed — Met Protocol-defined Stopping Criteria | 9 | 13 | 24 | 15

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo QD via a DPI in the morning for 24 weeks.
- UMEC 62.5 µg QD: Participants received UMEC 62.5 µg QD via a DPI in the morning for 24 weeks.
- VI 25 µg QD: Participants received VI 25 µg QD via a DPI for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | Total
Number analyzed (Participants) | 280 | 418 | 421 | 413 | 1532
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (9.04) | 64.0 (9.16) | 62.7 (8.52) | 63.1 (8.71) | 63.1 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 120 | 136 | 108 | 449
  Male | 195 | 298 | 285 | 305 | 1083
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 9 | 14 | 9 | 15 | 47
  American Indian or Alaska Native | 1 | 3 | 5 | 0 | 9
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 1 | 2
  Asian - East Asian Heritage | 1 | 2 | 2 | 1 | 6
  Asian - Japanese Heritage | 12 | 18 | 18 | 20 | 68
  Asian - South East Asian Heritage | 9 | 15 | 13 | 13 | 50
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 237 | 354 | 363 | 348 | 1302
  White - Mixed Race | 0 | 0 | 1 | 0 | 1
  Mixed Race | 11 | 12 | 9 | 14 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) on Day 169 (Week 24)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84, 112, 168, and 169. Baseline is defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Trough FEV1 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after the previous morning's dosing (ie., trough FEV1 on Day 169 is the mean of the FEV1 values obtained 23 and 24 hours after the morning dosing on Day 168). Change from Baseline at a particular visit was calculated as the trough FEV1 at that visit minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline , smoking status, center group, day, and day by Baseline and day by treatment interactions. ITT=Intent-to-Treat; par.=participants.
Time Frame: Baseline and Day 169
Population: Intent-to-Treat (ITT) Population: all par. randomized to trt. who received at least one dose of randomized study drug. Par. represents those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD
Number analyzed (Participants) | 201 | 322 | 317 | 330
Liters | 0.004 (0.0158) | 0.119 (0.0126) | 0.076 (0.0127) | 0.171 (0.0126)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.115, 95% CI 2-sided [0.076 to 0.155] — Least squares mean difference=UMEC 62.5 µg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs VI 25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.072, 95% CI 2-sided [0.032 to 0.112] — Least squares mean difference=VI 25 µg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.167, 95% CI 2-sided [0.128 to 0.207] — Least squares mean difference=UMEC/VI 62.5/25 µg minus Placebo
Statistical Analysis 4: Comparison: UMEC 62.5 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.052, 95% CI 2-sided [0.017 to 0.087] — Least squares mean difference=UMEC/VI 62.5/25 minus UMEC 62.5 µg
Statistical Analysis 5: Comparison: VI 25 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.095, 95% CI 2-sided [0.060 to 0.130] — Least squares mean difference=UMEC/VI 62.5/25 minus VI 25 µg

2. Secondary Outcome: Mean Transition Dyspnea Index (TDI) Focal Score at Day 168 (Week 24)
Description: Considered an 'other' endpoint by the FDA. The TDI is an interviewer-administered instrument which measures the changes in the participant's dyspnea from Baseline. This questionnaire was collected on Days 28, 84 and 168. The scores in the TDI evaluate ratings for 3 different categories (functional impairment, magnitude of task in exertional capacity, and magnitude of effort). TDI scores ranged from -3 (major deterioration) to +3 (major improvement); total score = -9 to 9. Analysis was performed using a repeated measures model with covariates of treatment, Baseline dyspnea index (BDI) focal score,smoking status, center group, day, day by BDI focal score and day by treatment interactions.
Time Frame: Day 168 (Week 24)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD
Number analyzed (Participants) | 204 | 326 | 317 | 336
Scores on a scale | 1.2 (0.20) | 2.2 (0.16) | 2.1 (0.16) | 2.4 (0.16)

3. Secondary Outcome: Change From Baseline in Weighted Mean (WM) 0-6 Hour FEV1 Obtained Post-dose at Day 168
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated at Days 1, 28, 84, and 168 using the 0-6-hour post-dose FEV1 measurements collected on that day, which included pre-dose (Day 1: 30 minutes [min] and 5 min prior to dosing; other serial visits: 23 and 24 hours after the previous morning dose) and post-dose at 15 min, 30 min, 1 hour, 3 hours, and 6 hours. Change from Baseline at a particular visit was calculated as the WM at that visit minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the two assessments made 30 min and 5 min pre-dose on Day 1), smoking status, center group, day, and day by Baseline and day by treatment interactions.
Time Frame: Baseline and Day 168
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD
Number analyzed (Participants) | 206 | 319 | 311 | 333
Liters | 0.001 (0.0158) | 0.151 (0.0128) | 0.123 (0.0128) | 0.243 (0.0127)

4. Other Pre Specified Outcome: Change From Baseline in the Mean Shortness of Breath With Daily Activities (SOBDA) Score for Week 24
Description: The newly developed SOBDA questionnaire assesses dyspnea or shortness of breath (SOB) with daily activities. The SOBDA questionnaire is made up of 13 items completed by the participant (par.) each evening prior to bedtime, when the par. is instructed to reflect on the current day's activities. The daily score is computed as the mean of the scores on the 13 items (>=7 items must have non-missing responses for this to be calculated). The par. is assigned a weekly mean SOBDA score ranging from 1 to 4 (greater scores indicate more severe breathlessness with daily activities) based on the mean of 7 days of data (>=4 of 7 days must be completed for a weekly mean to be calculated). Change from BL is the mean weekly SOBDA score minus BL. Analysis was performed using MMRM with covariates of treatment, BL (mean score in the week prior to treatment), smoking status, center group, week, week by BL and week by treatment interactions. This MMRM analysis only included Weeks 4, 8, 12, and 24.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD
Number analyzed (Participants) | 125 | 209 | 202 | 230
Scores on a scale | -0.06 (0.037) | -0.16 (0.029) | -0.21 (0.030) | -0.23 (0.029)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to 24 weeks).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants who had received at least one dose of randomized study medication during treatment period.
Arm/Group | Placebo | UMEC 62.5 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD
Serious Adverse Events (participants affected / at risk) | 9/280 | 27/418 | 24/421 | 21/413
Other Adverse Events (participants affected / at risk) | 62/280 | 96/418 | 87/421 | 93/413
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=280) | UMEC 62.5 µg QD (N=418) | VI 25 µg QD (N=421) | UMEC/VI 62.5/25 µg QD (N=413)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 8 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Infective exacerbation of chronic obstructive airway disease (Infections and infestations) | 0 | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2 | 0
Encephalitis (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=280) | UMEC 62.5 µg QD (N=418) | VI 25 µg QD (N=421) | UMEC/VI 62.5/25 µg QD (N=413)
Nasopharyngitis (Infections and infestations) | 16 | 29 | 26 | 39
Upper respiratory tract infection (Infections and infestations) | 14 | 21 | 17 | 13
Headache (Nervous system disorders) | 26 | 32 | 25 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 15 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 14 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 7 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.